CLINICAL TRIAL: NCT06970184
Title: Alveolar Ridge Preservation With Cortico-cancellous Collagenic Porcine Bone
Brief Title: Alveolar Ridge Preservation With Cortico-cancellous Porcine Bone
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Full Professor, University of Pisa
Other Study IDs: BONEISTO_ARP
Record Dates: First submitted 2025-04-23; First posted 2025-05-14 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Alveolar Ridge Preservation; Implant Therapy; Tooth Extraction Site Healing
Keywords: ARP; tooth extraction; dental implants; porcine bone; collagen
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARP 50:50: Tooth extraction + ARP with collagenated porcine bone hand-mixed (ratio 50:50) with a thermogel
  Interventions: Procedure: tooth extraction with alveolar ridge preservation; Procedure: Implant placement
- ARP 80:20: Tooth extraction + ARP with collagenated porcine bone pre-mixed (ratio 80:20) with a thermogel
  Interventions: Procedure: tooth extraction with alveolar ridge preservation; Procedure: Implant placement

INTERVENTIONS:
Procedure: tooth extraction with alveolar ridge preservation — alveolar ridge preservation performed after tooth extraction
Procedure: Implant placement — Implant placement

SUMMARY:
Observational, prospective study conducted on patients requiring tooth extractions followed by ARP and subsequent implant placement.

DETAILED DESCRIPTION:
The primary aim of this study is to compare the histomorphometric characteristics of two different formulations of CCPB used for ARP, and the secondary aim is to evaluate and compare clinical and aesthetic outcomes of dental implants placed in augmented sites.

Patients requiring the extraction of an hopeless tooth followed by ARP and subsequent implant placement are considered potentially eligible for the study.

At T0, Tooth extractions are performed trying to reduce the surgical trauma as possible. ARP is performed with 2 different combinations of a cortico-cancellous porcine bone with a thermogel (50:50 ratio, hand-mixed or 80:20 ratio, pre-mixed).

After 4 months of healing, patients undergo a radiographic examination before implant placement.

A T1, Implant site preparation is carried out using a trephine bur (to remove a core biopsy of the bone) followed by conventional osteotomy drills, and bone-level implants are placed. Bone samples are analyzed to evaluate new bone formation, presence of residual graft particles and marrow spaces.

Three months after placement, all implants are rehabilitated with screw-retained prosthetic crowns (T2).

Follow up is scheduled 1 year after prosthetic loading (T3).

ELIGIBILITY:
Inclusion Criteria:

* 18 yo
* Needing tooth extraction followed by ARP and implant-prosthetic rehabilitation

Exclusion Criteria:

* uncontrolled systemic diseases
* uncontrolled periodontitis
* undergoing previous or actual treatment with medications/radiations potentially impairing hard and soft tissues healing
* women during pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring hopeless tooth extraction followed by ARP and implant-prosthetic rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric characteristics of the bone: Newly formed bone (NB) | T1= 4 months following tooth extraction + ARP
  The primary outcome is evaluated in terms of Percentages of newly formed bone (NB) in the in the histological samples.
Histomorphometric characteristics of the bone: marrow spaces (MS) | T1= 4 months following tooth extraction + ARP
  The primary outcome is evaluated in terms of Percentages of marrow spaces (MS) in the histological samples
Histomorphometric characteristics of the bone: residual graft particles (RP) | T1= 4 months following tooth extraction + ARP
  The primary outcome is evaluated in terms of Percentages of marrow spaces (MS) in the histological samples

SECONDARY OUTCOMES:
Marginal Bone Level | T1= 4 months following tooth extraction + ARP
  Radiographic marginal bone level (measured in millimeters) taken at the mesial and distal aspect of the implant as the distance from the implant-abutment interface to the most apical bone-implant contact.
Marginal Bone Level | T2= 3 months following implant placement
  Radiographic marginal bone level (measured in millimeters) taken at the mesial and distal aspect of the implant as the distance from the implant-abutment interface to the most apical bone-implant contact.
Marginal Bone Level | T3= 1-year follow-up
  Radiographic marginal bone level (measured in millimeters) taken at the mesial and distal aspect of the implant as the distance from the implant-abutment interface to the most apical bone-implant contact.
Horizontal alveolar measure | Day 1 = tooth extraction + ARP
  Maximum post-extractive buccal/lingual distance (measured in millimeters) of the socket evaluated with a UNC periodontal probe
Horizontal alveolar measure | T1= 4 months following tooth extraction + ARP
  Maximum alveolar crest width at implant placement (measured in millimeters) evaluated with a UNC periodontal probe
Vertical alveolar measure | Day 1 = tooth extraction + ARP
  Mean distance (measured in millimeters) between mesial and distal reference points and the alveolar crest measured with a UNC periodontal probe
Vertical alveolar measure | T1= 4 months following tooth extraction + ARP
  Mean distance (measured in millimeters) between mesial and distal reference points and the alveolar crest measured with a UNC periodontal probe
Aesthetic outcomes | T2= 3 months following implant placement
  evaluated with the Pink Esthetic Score (PES) according to seven variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar ridge deficiency, soft tissue color, and soft tissue texture. Each variable could have a score ranging between 0 to 2; the total PES has a maximum level of 14
Aesthetic outcomes | T3= 1-year follow-up
  evaluated with the Pink Esthetic Score (PES) according to seven variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar ridge deficiency, soft tissue color, and soft tissue texture. Each variable could have a score ranging between 0 to 2; the total PES has a maximum level of 14

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Odontostomatologia e Chirurgia del Cavo Orale, Pisa, Italy, Italy

IPD SHARING:
Plan to Share IPD: No